CLINICAL TRIAL: NCT02371473
Title: Effect of Acetazolamide on Central Sleep Apnea Related to Opium Consumption
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Collaborators: Masih Daneshvari Hospital (Other)
Responsible Party: Principal Investigator, Parisa Adimi, Associate Professor of Medicine, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CRD-93-04
Record Dates: First submitted 2014-12-06; First posted 2015-02-25 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Central Sleep Apnea, Secondary
Keywords: Acetazolamide; Central Sleep Apnea; Opium Abuse
MeSH Terms: conditions — Sleep Apnea, Central; Opium Dependence

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- #1 (Acetazolamide-placebo) (Experimental): The arm #1 consists of 6 eligible patients who receive Acetazolamide 250mg once daily an hour before sleep for first six nights and after two weeks washout they receive placebo for six nights in the same order. After each six-day period they undergo polysomnography.
  Interventions: Drug: Acetazolamide-placebo
- #2 (Placebo-acetazolamide) (Experimental): The arm #2 consists of 6 eligible patients who receive placebo once daily an hour before sleep for first six nights and after two weeks washout they receive acetazolamide 250mg for six nights in the same order. After each six-day period they undergo polysomnography.
  Interventions: Drug: Placebo-acetazolamide

INTERVENTIONS:
Drug: Acetazolamide-placebo — The patients in this arm are given Acetazolamide mg for six days and after 2 weeks washout they are given placebo for six days.
  Other Names: Diamox. Drug and placebo are prepared in similar capsules.
  Arms: #1 (Acetazolamide-placebo)
Drug: Placebo-acetazolamide — The patients in this arm are given placebo for six days and after 2 weeks washout they are given Acetazolamide for six days.
  Other Names: Diamox. Drug and placebo are prepared in similar capsules.
  Arms: #2 (Placebo-acetazolamide)

SUMMARY:
Acetazolamide improves central sleep apnea related to opium consumption.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled, cross-over designed study to evaluate the effect of acetazolamide on central apneas in opium-user patients.

We are going to invite 12 eligible patients to enter our study. this sample will be obtained from the referral patients to Masih Daneshvari hospital sleep Lab. Eligible patients will undergo a full night polysomnography (PSG) to have a new measure of apnea indexes as baseline. Epwoth Sleepiness Scale Questionnaire (ESS) will be filled by the patient the night of the study.also an arterial blood sample will be obtained at the morning of each study. if the patient have more than 5 central apneas in each hour he/she will be scheduled to randomly receive a box containing 6 capsules to use one hour before bedtime at coming nights. The prescriber physician who will also score the tests and the patients are unaware either these capsules are acetazolamide 250mg or placebo. at 6th night we will perform PSG together with ESS questionnaire and arterial blood gas (ABG). after 2 weeks washout the patient receive another box containing 6 capsules with similar appearance to previous ones. If the patient receives acetazolamide in the first six nights, he/she will receive placebo in the second phase of the study and if the patient receives placebo in the first phase, he/she will receive acetazolamide in the second phase.

after the second 6 days, the third PSG will be performed plus ESS measurement and morning ABG sampling. Coded polysomnograms will be scored blindly.

ELIGIBILITY:
Inclusion Criteria:

* Opium or opioid use for at least two months in a daily manner
* Presence of five or more central sleep apnea per hour in a full-night recorded PSG

Exclusion Criteria:

* Congestive heart failure
* living in high altitude
* Chronic Obstructive Pulmonary Disease (COPD)
* Carbon dioxide partial pressure (pCO2) elevation due to other respiratory diseases
* Body Mass Index (BMI) > 32
* Obesity Hypoventilation Syndrome
* Severe renal or liver disorders
* Using Benzodiazepine
* Using Theophylline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2014-11; Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Changes in Central Apnea Index | baseline and six days

SECONDARY OUTCOMES:
Changes in daytime sleepiness, as measured by Epworth Sleepiness Scale (0-24) | baseline and six days

CONTACTS AND LOCATIONS:
Overall Officials: Parisa Adimi, MD, Principal Investigator — Shahid Beheshti University of Medical Sciences; Moein Forughi, MD, Study Director — Shaheed Behesti Medical University
Locations (1):
- Masih Daneshvari Hospital, Tehran, Iran

REFERENCES:
- [Derived] Naghan PA, Raeisi K, Khoundabi B, Foroughi M, Malekmohammad M, Mohebbi M, Bagheri A, Fahimi F. The effect of acetazolamide on the improvement of central apnea caused by abusing opioid drugs in the clinical trial. Sleep Breath. 2020 Dec;24(4):1417-1425. doi: 10.1007/s11325-019-01968-3. Epub 2019 Dec 5. PMID 31808012